CLINICAL TRIAL: NCT01611701
Title: Cryoballoon Ablation of Pulmonary Veins After Failed Radiofrequency Ablation in Patients With Paroxysmal Atrial Fibrillation
Brief Title: Cryoballoon Ablation of Pulmonary Veins After Failed RF Ablation in Patients With Paroxysmal AF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RFA-655-CA
Record Dates: First submitted 2012-05-25; First posted 2012-06-05 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cryoballoon group (Active Comparator)
  Interventions: Procedure: cryoballoon ablation
- RF group (Active Comparator)
  Interventions: Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: cryoballoon ablation — In Cryo group, 28mm balloon was introduced into the PV ostium with the best possible occlusion of the PV. Every step was controlled by fluoroscopy. Cryoenergy was applied for maximal 6 minutes per application for 2 times, resulting in a circumferential ablation lesion. Before the right superior vein was treated, a quadripolar catheter was placed in the superior vena cava to continuously stimulate the right phrenic nerve during cryoapplication. The application was stopped immediately in the case of diminished diaphragm movements.
  Arms: Cryoballoon group
Procedure: Radiofrequency ablation — n RF group, reisolation of the PV was performed by identifying the breakthrough site. Radiofrequency energy was delivered at 43°C, 35 W, 0.5 cm away from the PV ostia at the anterior wall, and was reduced to 43°C, 30 W, 1 cm away from the PV ostia at the posterior wall, with a saline irrigation rate of 17 mL/min. Each lesion was ablated continuously until the local potential amplitude decreased by >80% or RF energy deliveries exceeded 40 s.
  Arms: RF group

SUMMARY:
The aim of this prospective randomized double-blind study was to compare the efficacy and safety of cryoballoon ablation with the RF approach in the treatment of paroxysmal AF after failed first radiofrequency ablation.

ELIGIBILITY:
Inclusion Criteria:

* Previous failed first radiofrequency ablation procedure (only circumferential PV isolation without linear lesions) in patients referred for second catheter ablation of AF
* > 3 months after first PVI

Exclusion Criteria:

* Congestive heart failure
* Ejection fraction <35%
* Left atrial diameter >60 mm

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-10; Primary Completion 2011-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Recurrence of atrial tachyarrhythmia, including AF and left atrial flutter/tachycardia, after a second ablation procedure | 1 year

SECONDARY OUTCOMES:
Percentage of complication after procedure between two groups | 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- The Valley Health System and Columbia University College of Physicians & Surgeons, New York, New York, United States
- State Research Institute of Circulation Pathology, Novosibirsk, Russia

REFERENCES:
- [Derived] Pokushalov E, Romanov A, Artyomenko S, Baranova V, Losik D, Bairamova S, Karaskov A, Mittal S, Steinberg JS. Cryoballoon versus radiofrequency for pulmonary vein re-isolation after a failed initial ablation procedure in patients with paroxysmal atrial fibrillation. J Cardiovasc Electrophysiol. 2013 Mar;24(3):274-9. doi: 10.1111/jce.12038. Epub 2012 Dec 4. PMID 23210695
- See also: State Research Institute of Circulation Pathology Official Site — http://meshalkin.ru